CLINICAL TRIAL: NCT01256320
Title: The Impact of Egg Consumption on Indices of Vascular Health in Individuals With Peripheral Arterial Disease
Brief Title: Egg Study With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. J. House, Professor and Head, Deparment of Human Nutritional Sciences, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H2009:081:110
Record Dates: First submitted 2010-06-18; First posted 2010-12-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): no shell egg consumption and usual dietary practices
- Classic Egg Group (Active Comparator): consumption of 6 eggs/week (1 egg/day for 6 days with 1 day rest) of commercial classic eggs
  Interventions: Other: Classic Egg Group
- Omega 3 Egg Group (Active Comparator): consumption of 6 eggs/week (1 egg/day for 6 days with 1 day rest) of commercial Omega-3 eggs
  Interventions: Other: Omega 3 Egg Group

INTERVENTIONS:
Other: Classic Egg Group — consumption of 6 eggs/week (1 egg/day for 6 days with 1 day rest) of commercial classic eggs
  Arms: Classic Egg Group
Other: Omega 3 Egg Group — consumption of 6 eggs/week (1 egg/day for 6 days with 1 day rest) of commercial Omega-3 eggs
  Arms: Omega 3 Egg Group

SUMMARY:
The current research study has the potential to generate data that would provide solid clinical endpoints as to the impact of including eggs in a regular diet in individuals with peripheral arterial disease. Any one of three potential outcomes may be observed as a result of this study, and they are predicted as follows: 1) Egg consumption does not lead to a deterioration of indices of cardiovascular health; 2) Egg consumption improves indices of cardiovascular health; 3) Egg consumption worsens the indices of cardiovascular health.

DETAILED DESCRIPTION:
Given the hypotheses proposed, if either of the first two predictions prove to be positive, they will help encourage directive efforts to be made toward effective nutrition messages for egg consumption in the peripheral arterial disease and the healthy population. If the last prediction is positive, while least favourable, it will still establish important information to assist the industry in their efforts toward establishing population-specific nutrition messaging.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of peripheral arterial disease including those with claudication as defined by an ankle brachial index of ≤ 0.90 or asymptomatic carotid stenosis of > 50%; or who have had a previous intervention for peripheral arterial disease;
2. Male or female, > 40 years of age;
3. Willing to comply with the protocol requirements;
4. Willing to provide informed consent;
5. Stable medication profile with no changes anticipated for the duration of the proposed study schedule (8 weeks);
6. Participants having completed the Flax Study are eligible to participate if their completion has been more than 3 months.

Exclusion Criteria:

1. Renal failure requiring dialysis;
2. Diabetes, requiring diabetic medication; Participants with diabetes who do not require diabetic medication and have good glycemic control will be eligible for participation in the study. Participant with elevated fasting blood glucose levels and glycated hemoglobin above 'standard of care' at baseline will not proceed with the study;
3. Hyperlipidemia as defined by a cholesterol of >4.1 mmol/L (as per the National Cholesterol Education Program Adult Treatment Panel III, (NCEP ATP III) guidelines;
4. Hormone replacement therapy;
5. Inability to adhere to a regular diet;
6. Habitual egg intake of 5 or more eggs per week;
7. History of gastrointestinal reactions or allergies to eggs;
8. Daily consumption of omega-3 supplements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Establish quantitative and qualitative data on the dietary patterns, including egg consumption, in patients with PAD | change in assessments from baseline to 8 weeks
  The following assessments are included to measure the primary outcome:
  1)Anthropometrics: weight, height; waist circumference, Body Mass Index; 2)Dietary Assessment:3-day dietary food record, food frequency questionnaire (baseline only); 3)Biochemical Analyses; 4)Expression and Metabolic Profiling; 5)Arterial Compliance: Ankle-brachial index, pulse wave velocity, arterial vasodilation, and advanced glycation endproducts; 6) Semi-structured interview.

SECONDARY OUTCOMES:
Determine the impact of consuming 6 eggs per week on primary end-points and other modifiable risk factors in patients with PAD. | change in assessments from baseline to 8 weeks
  The following assessments are included to measure the primary outcome:
  1)Anthropometrics: weight, height; waist circumference, Body Mass Index; 2)Dietary Assessment:3-day dietary food record, food frequency questionnaire (baseline only); 3)Biochemical Analyses; 4)Expression and Metabolic Profiling; 5)Arterial Compliance: Ankle-brachial index, pulse wave velocity, arterial vasodilation, and advanced glycation endproducts; 6) Semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: James House, PhD, Principal Investigator — University of Manitoba
Locations (1):
- IH Asper Clinical Research Institute, St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Calabro P, Yeh ET. The pleiotropic effects of statins. Curr Opin Cardiol. 2005 Nov;20(6):541-6. doi: 10.1097/01.hco.0000181482.99067.bf. PMID 16234628
- [Background] Eberhardt RT, Coffman JD. Cardiovascular morbidity and mortality in peripheral arterial disease. Curr Drug Targets Cardiovasc Haematol Disord. 2004 Sep;4(3):209-17. doi: 10.2174/1568006043336230. PMID 15379611
- [Background] Ismail HM, Jackson K, Smith D. Diagnosis and treatment of peripheral arterial disease compared with other atherosclerotic vascular diseases in a university primary care clinic. J Investig Med. 2006 Jul;54(5):255-61. doi: 10.2310/6650.2006.05049. PMID 16984798
- [Background] Katz DL, Evans MA, Nawaz H, Njike VY, Chan W, Comerford BP, Hoxley ML. Egg consumption and endothelial function: a randomized controlled crossover trial. Int J Cardiol. 2005 Mar 10;99(1):65-70. doi: 10.1016/j.ijcard.2003.11.028. PMID 15721501
- [Background] Kressel G, Trunz B, Bub A, Hulsmann O, Wolters M, Lichtinghagen R, Stichtenoth DO, Hahn A. Systemic and vascular markers of inflammation in relation to metabolic syndrome and insulin resistance in adults with elevated atherosclerosis risk. Atherosclerosis. 2009 Jan;202(1):263-71. doi: 10.1016/j.atherosclerosis.2008.04.012. Epub 2008 Apr 20. PMID 18501910
- [Background] Lahera V, Goicoechea M, de Vinuesa SG, Miana M, de las Heras N, Cachofeiro V, Luno J. Endothelial dysfunction, oxidative stress and inflammation in atherosclerosis: beneficial effects of statins. Curr Med Chem. 2007;14(2):243-8. doi: 10.2174/092986707779313381. PMID 17266583
- [Background] Lane JS, Magno CP, Lane KT, Chan T, Hoyt DB, Greenfield S. Nutrition impacts the prevalence of peripheral arterial disease in the United States. J Vasc Surg. 2008 Oct;48(4):897-904. doi: 10.1016/j.jvs.2008.05.014. Epub 2008 Jun 30. PMID 18586439
- [Background] Third Report of the National Cholesterol Education Program (NCEP) on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel, ATP III) 2001; U.S. Department of Health & Human Services
- [Background] Raitakari et al. 2008 Br J Nutr 18:1
- [Background] Ratliff JC, Mutungi G, Puglisi MJ, Volek JS, Fernandez ML. Eggs modulate the inflammatory response to carbohydrate restricted diets in overweight men. Nutr Metab (Lond). 2008 Feb 20;5:6. doi: 10.1186/1743-7075-5-6. PMID 18289377
- [Background] Shuaibi et al. 2008a; Journal of the American Dietetic Association, In Press
- [Background] Shuaibi et al. 2008b; Journal of the American Dietetic Association, In Press
- [Background] Weatherley BD, Nelson JJ, Heiss G, Chambless LE, Sharrett AR, Nieto FJ, Folsom AR, Rosamond WD. The association of the ankle-brachial index with incident coronary heart disease: the Atherosclerosis Risk In Communities (ARIC) study, 1987-2001. BMC Cardiovasc Disord. 2007 Jan 16;7:3. doi: 10.1186/1471-2261-7-3. PMID 17227586
- [Background] Weingartner O, Lutjohann D, Ji S, Weisshoff N, List F, Sudhop T, von Bergmann K, Gertz K, Konig J, Schafers HJ, Endres M, Bohm M, Laufs U. Vascular effects of diet supplementation with plant sterols. J Am Coll Cardiol. 2008 Apr 22;51(16):1553-61. doi: 10.1016/j.jacc.2007.09.074. PMID 18420097